CLINICAL TRIAL: NCT01751399
Title: A Single Dose Pharmacokinetic Study of LY2605541 in Subjects With Hepatic Impairment
Brief Title: A Single Dose Study of LY2605541 in Participants With Liver Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14205; I2R-MC-BIDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers; Hepatic Insufficiency; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hepatic Insufficiency; Diabetes Mellitus, Type 2 | interventions — LY2605541

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2605541-Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive a single subcutaneous (SC) dose of 0.075 milligrams per kilogram (mg/kg) LY2605541
  Interventions: Drug: LY2605541
- LY2605541-Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment will receive a single SC dose of 0.075 mg/kg LY2605541
  Interventions: Drug: LY2605541
- LY2605541-Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment will receive a single SC dose of 0.075 mg/kg LY2605541
  Interventions: Drug: LY2605541
- LY2605541-Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment will receive a single SC dose of 0.075 mg/kg LY2605541
  Interventions: Drug: LY2605541

INTERVENTIONS:
Drug: LY2605541

SUMMARY:
The primary purpose of this study is to help answer the following research questions:

* To evaluate how much of the study drug (LY2605541) is in the blood of participants with varying degrees of liver impairment compared to those with normal liver function
* To assess the safety of LY2605541 and any side effects that might be associated with it

DETAILED DESCRIPTION:
The study is conducted in 4 groups, based on the Child-Pugh classification of hepatic impairment as follows:

Group 1: Participants with normal hepatic function (Control); Group 2: Participants with mild hepatic impairment (Child-Pugh class A); Group 3: Participants with moderate hepatic impairment (Child-Pugh class B); and Group 4: Participants with severe hepatic impairment (Child-Pugh class C).

ELIGIBILITY:
Inclusion Criteria:

All Participants (including those with type 2 diabetes mellitus [T2DM] who are controlled by diet)

* Male participants agree to use a reliable method of birth control during the study
* Female participants of child-bearing potential (not surgically sterilized between menarche and menopause) must have a negative pregnancy test at the time of enrollment and must be using a reliable method of birth control
* Women of non-child-bearing potential due to surgical sterilization (at least 6 weeks after surgical bilateral oophorectomy with or without hysterectomy or at least 6 weeks after tubal ligation) confirmed by medical history, or menopause.
* Menopausal women include women with either spontaneous amenorrhea for at least 12 months or spontaneous amenorrhea for 6 to 12 months and a follicle-stimulating hormone (FSH) level greater than 40 milli international units per milliliter (mIU/mL)
* Have a body mass index (BMI) of 18.5 to 40 kilogram per square meter (kg/m^2)
* Have normal sitting blood pressure and heart rate compatible with their disease state
* Have venous access sufficient to allow blood sampling
* Have given written informed consent approved by Lilly and the Ethical Review Board (ERB) governing the site

Participants with Normal Hepatic Function

* Overtly healthy males or females with normal hepatic function
* Have clinical laboratory test results within normal reference range for the investigator site, or results with minor deviations not considered to be clinically significant by the investigator

Participants with Hepatic Impairment

* Have stable liver impairment with no sign of recent deterioration (alcoholic, posthepatitis, biliary cirrhosis, or cryptogenic) classified as Child-Pugh class A, B, or C who are considered by the investigator as acceptable for participation in the study

Exclusion Criteria:

All Participants (including those with T2DM)

* Are currently enrolled in, have completed or discontinued within the last 30 days from a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have an acute infection with fever or infectious disease or febrile illness within 3 days prior to administration of the study medication
* Have known allergies or significant hypersensitivity to LY2605541, its excipients, or related compounds, or history of relevant allergic reactions of any origin
* Have previously completed or withdrawn from this study or any other study investigating LY2605541 and have previously received the investigational product
* Have Type 1 Diabetes Mellitus (T1DM) or have T2DM and are receiving anti-diabetic medication
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have had a liver transplant or have taken immunosuppressants following any organ transplant
* Have shown signs of variceal bleeding during the last 2 weeks prior to screening
* Show evidence of irritable bowel syndrome, chronic diarrhea, other symptomatic digestive problems or a known history of repeated chronic stool positive for occult blood, or be considered by the investigator to be at greater risk of acute or chronic pancreatitis
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to stop alcohol consumption for the duration of the study (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Are on total parenteral nutrition
* Take anticoagulants for therapeutic use, other than low dose acetylsalicyclic acid
* Are excessive consumers of xanthines

Participants with Normal Hepatic Function

* Have any medically significant history of neurologic disease, cancer, or cardiac, respiratory, metabolic, hepatic, renal, gastrointestinal (except appendectomy and cholecystectomy), dermatological, venereal, hematological disorder or disease
* Have creatinine clearance (CrCl) less than 80 milliliters per minute (mL/min)
* Show evidence of significant active neuropsychiatric disease in the opinion of the investigator
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Show evidence of hepatitis C and/or positive hepatitis C antibody

Participants with Hepatic Impairment

* Show evidence of any significant active disease other than that responsible for or associated with mild, moderate, or severe hepatic impairment
* Show evidence of hepatorenal syndrome as shown by CrCl <50 mL/min calculated using the Cockcroft-Gault equation
* Have shown signs of spontaneous bacterial peritonitis within 6 months prior to enrollment into the study
* Have severe hyponatremia (sodium <120 millimoles per liter [mmol/L])
* Show signs of hepatocellular carcinoma
* Have a portal shunt
* Show, in the opinion of the investigator, evidence of significant active neuropsychiatric disease other than grade 1 hepatic encephalopathy
* Have hemoglobin concentrations <9.0 grams per deciliter (g/dL)
* Have a platelet count of <30 x 10^9 cells per liter (cells/L), unless, after consultation with the sponsor, they are considered as acceptable for participation in the study
* Have total serum bilirubin concentrations >15 milligrams per deciliter (mg/dL) (>257 micromoles per liter [μmol/L])
* Take medications known to interfere with hepatic metabolism (for example barbiturates or phenothiayines) or known to alter other major organ systems
* Show signs of acute cholestasis or acute cholecystitis
* Have severe ascites

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Balatonfüred, Hungary

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2605541-Normal Hepatic Function: Participants with normal hepatic function received a single subcutaneous (SC) dose of 0.075 milligrams per kilogram (mg/kg) LY2605541
- LY2605541-Mild Hepatic Impairment: Participants with mild hepatic impairment received a single SC dose of 0.075 mg/kg LY2605541
- LY2605541-Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single SC dose of 0.075 mg/kg LY2605541
- LY2605541-Severe Hepatic Impairment: Participants with severe hepatic impairment received a single SC dose of 0.075 mg/kg LY2605541
Period: Overall Study
Arm/Group | LY2605541-Normal Hepatic Function | LY2605541-Mild Hepatic Impairment | LY2605541-Moderate Hepatic Impairment | LY2605541-Severe Hepatic Impairment
Started | 12 | 8 | 8 | 7
Received 1 Dose of Study Drug | 12 | 8 | 8 | 7
Completed | 12 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- LY2605541-Normal Hepatic Function: Participants with normal hepatic function received a single SC dose of 0.075 mg/kg LY2605541
- Total: Total of all reporting groups
Arm/Group | LY2605541-Normal Hepatic Function | LY2605541-Mild Hepatic Impairment | LY2605541-Moderate Hepatic Impairment | LY2605541-Severe Hepatic Impairment | Total
Number analyzed (Participants) | 12 | 8 | 8 | 7 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (6.4) | 56.0 (5.9) | 52.4 (9.9) | 57.6 (3.3) | 54.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 3 | 3 | 15
  Male | 6 | 5 | 5 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 8 | 8 | 7 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 12 | 8 | 8 | 7 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 5 | 4 | 4 | 5 | 18
  Germany | 7 | 4 | 4 | 2 | 17
Participants with Diabetes [Count of Participants; unit: Participants] | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve From Zero to Infinity (AUC[0-∞]) of LY2605541
Time Frame: Predose and 2, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours postdose
Population: All participants who received 1 dose of LY2605541 and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole*hours/liter (pmol*h/L)
Arm/Group | LY2605541-Normal Hepatic Function | LY2605541-Mild Hepatic Impairment | LY2605541-Moderate Hepatic Impairment | LY2605541-Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 7
picomole*hours/liter (pmol*h/L) | 85200 (19) | 67200 (31) | 64300 (65) | 66600 (77)

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2605541
Time Frame: Predose and 2, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours postdose
Population: All participants who received 1 dose of LY2605541 and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | LY2605541-Normal Hepatic Function | LY2605541-Mild Hepatic Impairment | LY2605541-Moderate Hepatic Impairment | LY2605541-Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 7
pmol/L | 1300 (38) | 946 (73) | 1180 (163) | 1090 (119)

ADVERSE EVENTS:
Arm/Group | LY2605541-Normal Hepatic Function | LY2605541-Mild Hepatic Impairment | LY2605541-Moderate Hepatic Impairment | LY2605541-Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 5/12 | 1/8 | 1/8 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541-Normal Hepatic Function (N=12) | LY2605541-Mild Hepatic Impairment (N=8) | LY2605541-Moderate Hepatic Impairment (N=8) | LY2605541-Severe Hepatic Impairment (N=7)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days